CLINICAL TRIAL: NCT04065854
Title: Promoting Activity, Independence and Stability in Early Dementia and Mild Cognitive Impairment
Acronym: PrAISED2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17HC006
Record Dates: First submitted 2019-05-21; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Multi-centre, pragmatic, parallel-group, randomised controlled trial, with internal pilot trial, and embedded process and economic evaluations.
  Web-based randomisation, using a dynamic adaptive algorithm, stratified for centre and other variables to 1) active intervention or 2) standard brief falls assessment and advice. An internal pilot trial will recruit the first 50 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive standard brief falls assessment and advice.
- Intervention (Active Comparator): Therapy intervention.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Assessment, tailored strength and balance exercise programme, activity analysis and risk enablement advice, and assessment for environmental hazards. Tailored adherence support and supervision.
  Arms: Intervention

SUMMARY:
A clinical trial to test the clinical and cost-effectiveness of a therapy intervention designed to promote activity and independence and reduce falls, amongst people with early dementia or mild cognitive impairment

DETAILED DESCRIPTION:
Background and study aims People with memory problems can struggle with everyday activities and may stop doing things they want to do. They are more prone to accidents and have a higher risk of falling. Occupational therapists can advise how to do daily activities more easily and safely. Physiotherapists can teach exercises which increase activity and improve balance, and may help maintain memory. There is little research on how to make these interventions work for with people with memory problems. The aim of this study is to compare an activity and exercise programme developed for people with memory problems to standard falls prevention assessment and advice.

Who can participate? Patients aged 65 or over with early dementia or memory problems, recruited from memory clinics or the 'Join Dementia Research' register

What does the study involve? Participants are randomly allocated to either the control group or the intervention group. The control group receive standard brief falls assessment and advice, and up to two further visits if required. The intervention group receive an assessment, tailored strength and balance exercise programme, activity analysis and risk enablement advice, and assessment for environmental hazards. The intervention is delivered over 1 year in participants' own homes, and is tailored to individual interests, abilities and need for supervision. Participants are encouraged to exercise by themselves or with family members between visits, and once the programme ends. Researchers visit at the start of the study and after 12 months to measure ability in activities of daily living, activity, quality of life, memory and health service use. Participants complete monthly falls diaries over 15 months. The researchers conduct interviews and video record some therapy sessions to help understand how the programme works in practice.

What are the possible benefits and risks of participating? Some participants may benefit from taking part in the intervention, as exercise is generally known to be beneficial to health and well-being, including benefits to heart, blood pressure, diabetes, joints, mood and daily life. These participants may find that they are better able to do their daily activities. All participants and their relatives may enjoy having the researchers coming to visit them in their house. Some people appreciate having the opportunity to contribute to the well-being of others through research.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 or over (no maximum)
2. Diagnosis of MCI or dementia (of any subtype, except Dementia with Lewy Bodies i.e. Parkinson's Disease Dementia)
3. Have a carer or friend who knows the participant well (at least one hour a week contact over the phone, internet, or in person), and is willing and able to act as an informant
4. Able to walk without human help
5. Able to communicate in English
6. Able to see, hear and have dexterity sufficiently to perform neuropsychological tests
7. Have capacity to give consent to participate, and consenting to do so

Exclusion Criteria:

1. Co-morbidity preventing participation (e.g. severe breathlessness, pain, psychosis, Parkinson's, Dementia with Lewy Bodies, or other severe neurological disease)
2. Unavailable over the next year (e.g. plans to relocate or go on a long holiday, or has a life expectancy of less than a year)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-03-13 (Estimated)

PRIMARY OUTCOMES:
Disability Assessment in Dementia (DAD) | 12 months
  Primary outcomes will be disability in Activities of Daily Living (Disability Assessment in Dementia, DAD) measured 12 months after randomisation. This is as recommended in a recent NIHR systematic review [Webster 2017].
  scale range is 0% to 100%. Where 0% = minimal functional ability and 100% maximal functional ability. Higher scores represent less disability in ADL and lower scores indicate more dysfunction. There are no subscales.
  "The total score is obtained by adding the rating for each question and converting this total score out of 100. The items rated as N/A are not considered for the total score. For example:
  A score of 33 on 40 (maximum score) converted out of 100 = 83% A score of 33 on 38 (max. score with 2 N/A) converted out of 100 = 87%
  This will result in a final score, a percentage which provides an appreciation of global function in ADL. Higher scores represent less disability in ADL while lower scores indicate more dysfunction."

SECONDARY OUTCOMES:
Nottingham Extended ADL Scale | 12 months
  Self-reported Activities of Daily Living (ADL) using the Nottingham Extended ADL Scale [Nouri and Lincoln 1980].
Falls Rate | 12 months
  Falls rate in months four-15 from randomisation (defined as 'unintentionally coming to rest on the ground or at a lower level, however caused', and ascertained by monthly diary)
Quality of Life | 12 months
  Quality of life (EQ5D3L and EQ5D5L proxy [EuroQol Group 1990]; DemQol and DemQol proxy, including Demqol-u weights [Smith 2005; Mulhern 2013])
Mood or 'Affect' | 12 months
  Mood or 'Affect' - Hospital Anxiety and Depression Scale (HADS [Zigmond and Snaith 1983]; Apathy Evaluation Scale - AES [Marin, Biedrzycki and Firinciogullari 1991])
Physical activity | 12 months
  Longitudinal Aging Study Amsterdam (LASA) physical activity questionnaire [Stel 2004], pedometers
Cognition | 12 months
  three scales from CANTAB [Cambridge Cognition, 2015]; Montreal Cognitive Assessment - MoCA [Nasreddine 2005], verbal fluency (from MoCA)
Time to first fall | 12 months
  Time to first fall (from diary)
Rate of fractures and injurious falls | 12 months
  Rate of fractures and injurious falls (from diary)
Rate of hospital and care home admissions, and days spent in hospital | 12 months
  Rate of hospital and care home admissions, and days spent in hospital (from diary, hospital administrative records)
Carer strain | 12 months
  Carer strain (Carergiver Strain Index [Robinson 1983]).
Carer health-related quality of life | 12 months
  Carer health-related quality of life (EQ5D-5L [EuroQol Group 1990])
Personality | 12 months
  Personality (Big Five Personality Inventory- short [BFI-10, Rammstedt and John 2007])

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Derbyshire Healthcare NHS Foundation Trust, Derby, Derbyshire
  - Lincolnshire Partnership NHS Foundation Trust, Lincoln, Lincolnshire
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham, Notts
  - RICE - Research Institute for the Care of Older People, Bath, Somerset

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PrAISED website — http://nottingham.ac.uk/praised/index.aspx